CLINICAL TRIAL: NCT01478646
Title: The Effect of Reflective Breathing Therapy Compared With Conventional Breathing Therapy on Dyspnoea and Activity in Patients With COPD III-IV
Brief Title: The Effect of Reflective Breathing Therapy Compared With Conventional Breathing Therapy in Patients With Chronic Obstructive Pulmonary Disease (COPD) III-IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: University of Osnabrueck (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician (department of pulmonology), Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAT 2011; KBerchtesgadener (Registry Identifier: KBerchtesgadener)
Record Dates: First submitted 2011-09-30; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: breathing therapy; reflective breathing therapy; COPD; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional breathing therapy (Experimental): first: conventional breathing therapy, second: reflectory breathing therapy
  Interventions: Other: conventional breathing therapy
- Reflectory breathing therapy (Experimental): first: reflectory breathing therapy second: conventional breathing therapy
  Interventions: Other: reflectory breathing therapy

INTERVENTIONS:
Other: conventional breathing therapy — duration: 60 minutes.
  Arms: Conventional breathing therapy
Other: reflectory breathing therapy — duration: 60 minutes.
  Arms: Reflectory breathing therapy

SUMMARY:
The purpose of this study is to determine whether different types of breathing therapies in patients with COPD III-IV decrease dyspnea and increase activity.

DETAILED DESCRIPTION:
In the treatment of COPD-Patients different kinds of breathing therapy techniques are used, but many of them are not reassessed yet.

Dyspnea is one of the predominant symptoms of COPD patients and has negative impacts on the activity of the patients. Dyspnea during exertion leads to avoiding activity and results in a deconditioning of muscles and of the cardiovascular system.

Thus breathing therapy techniques seem to be useful, which may lead to a decrease of dyspnea and an increase of activity.

The purpose of this study is to determine whether reflective breathing therapy is more effective on decreasing dyspnea and increasing activity than conventional breathing therapy.

ELIGIBILITY:
Inclusion Criteria:

* inpatient rehabilitation
* COPD (Gold stage III and IV)

Exclusion Criteria:

* severe exacerbation in the last four weeks
* acute infections
* fever
* neuritides
* severe osteoporosis
* skin disease
* manic depression

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in BORG-Scale | Change from pre (minute o) in BORG-scale at directly post intervention (minute 60)
  Instrument for self-reported dyspnea; modified BORG-scale ranges from 1 (no dyspnea) to 10 (maximum dyspnea).

SECONDARY OUTCOMES:
Change in residual volume | change from pre (minute 0) in residual volume at post (minute 60) intervention
  measured by a portable spirometry device

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Dr. med., Study Chair — Schön Klinik Berchtesgadener Land; Stella Seeberg, Principal Investigator — University of Osnabrueck
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau, Bavaria, Germany